CLINICAL TRIAL: NCT04538261
Title: Elevation of the Fetal Buttocks Prior to External Cephalic Version
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not recruiting at the rate we thought it would.
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1379199
Record Dates: First submitted 2020-08-17; First posted 2020-09-04 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-12

CONDITIONS: Breech Presentation; External Cephalic Version
Keywords: Breech; Version
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Intervention Model Description: Randomized trial using control and interventional arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigators and participants will not know whether participants have undergone inflation of the balloon device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Sham Comparator): Non-inflation of the balloon device
  Interventions: Device: Fetal Pillow insertion
- Intervention (Experimental): Inflation of the balloon device
  Interventions: Device: Fetal Pillow insertion

INTERVENTIONS:
Device: Fetal Pillow insertion — Inflation of balloon device used to elevate fetal buttocks prior to performing external cephalic version procedure

SUMMARY:
This is a prospective, randomized double-blind clinical trial evaluating the effect of a balloon device (Fetal Pillow) to elevate the fetal buttocks during external cephalic version procedures. Eligible study population: nulliparous pregnant women between 37-40 weeks estimated gestational age with a breech presenting fetus and no contraindications to external cephalic version.

DETAILED DESCRIPTION:
Patients meeting inclusion criteria will be offered participation in this study. After performing an obstetric sonogram to determine fetal position, amniotic fluid status, fetal weight and placental location, the patient will be randomized to either placement of the Fetal Pillow balloon device with sham inflation (control arm) or placement of the device with inflation (study arm).

The researcher will show the patient the device, open the sterile container, and insert the device into the vagina per manufacturer's guidelines for all patients in the study. All patients will mark a line on a 100mm VAS to assess pre-insertion and post-insertion pain. The study physician will then obtain the assistance of a certified nurse midwife to inflate the device or perform a sham inflation. In order for the physician investigator to remain blinded, the physician will leave the room during the time of the inflation/sham inflation. A certified nurse midwife previously trained to inflate the device will perform the inflation or sham inflation per randomization. The assisting midwife will inflate the device with 180 mL of saline for those patients randomized to inflation. This will occur under a sheet so that the patient is blinded to the randomization scheme. If the patient is randomized to no inflation, the midwife will perform a sham inflation, also under a sheet. All patients will mark a line on a 100mm VAS to assess post-inflation/sham inflation pain. The assisting midwife then leaves the room, and the study physician reenters the room and proceeds with the external cephalic version (ECV) procedure.

Regardless of randomization, at this point the ECV procedure proceeds using normal routine. The ECV will be attempted up to four times and VAS will be assessed after each attempt. Once completed, all patients will also mark a line on a 100mm VAS to assess post-ECV pain.

The research physician will then remove the Fetal Pillow. Regardless of randomization, the procedure is completed per the usual routine of fetal monitoring, assessing for rupture of membranes, labor or bleeding, discussing post-procedure care, then discharge home (or, less likely, admitting for either observation or delivery).

The researcher will fill out the ECV portion of the data collection form. Data are collected later for delivery outcomes and costs for the mother and neonate.

ELIGIBILITY:
Inclusion Criteria:

1. Women delivering at AdventHealth Orlando campus.
2. Breech presenting part as diagnosed by bedside sonography.
3. No prior deliveries >/= 20 weeks gestational age.
4. Pregnancy is between 37-40 weeks gestational age.
5. Live fetus.
6. Patient is >/= age 18.
7. Patient speaks English or Spanish as primary language.
8. Patient able to understand verbal and written consent

Exclusion Criteria:

1. Non-breech presentation (cephalic, transverse, oblique).
2. More than 1 fetus.
3. Cervical dilation of >/= 1cm.
4. Prior uterine incision.
5. Congenital uterine anomaly.
6. Body mass index more than 40 kg/m2.
7. Uterine fibroids causing soft tissue dystocia.
8. Extended fetal neck.
9. Oligohydramnios (4-quadrant amniotic fluid index </= 5cm).
10. Spontaneous rupture of membranes.
11. Any contraindication to vaginal delivery.
12. Intrauterine growth restriction (estimated fetal weight </= 10%ile).
13. Estimated fetal weight > /= 5,000 grams for non-diabetic patient or >/= 4,500 grams for patient with pre-existing or gestational diabetes, confirmed by ultrasound.
14. Fetal gastroschisis.
15. Fetal neural tube defect.
16. Severe-range preeclampsia.
17. Patient had regional anesthesia immediately prior to ECV.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Hill, MD, Principal Investigator — AdventHealth; Ariana Mora, Study Director — AdventHealth
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of research team.

REFERENCES:
- [Background] External Cephalic Version: ACOG Practice Bulletin, Number 221. Obstet Gynecol. 2020 May;135(5):e203-e212. doi: 10.1097/AOG.0000000000003837. PMID 32332415
- [Result] Seal SL, Dey A, Barman SC, Kamilya G, Mukherji J, Onwude JL. Randomized controlled trial of elevation of the fetal head with a fetal pillow during cesarean delivery at full cervical dilatation. Int J Gynaecol Obstet. 2016 May;133(2):178-82. doi: 10.1016/j.ijgo.2015.09.019. Epub 2016 Jan 15. PMID 26868074
- [Result] Hofmeyr GJ, Kulier R, West HM. External cephalic version for breech presentation at term. Cochrane Database Syst Rev. 2015 Apr 1;2015(4):CD000083. doi: 10.1002/14651858.CD000083.pub3. PMID 25828903
- [Result] Kok M, Cnossen J, Gravendeel L, van der Post J, Opmeer B, Mol BW. Clinical factors to predict the outcome of external cephalic version: a metaanalysis. Am J Obstet Gynecol. 2008 Dec;199(6):630.e1-7; discussion e1-5. doi: 10.1016/j.ajog.2008.03.008. Epub 2008 May 23. PMID 18456227
- [Result] Weiniger CF, Ginosar Y, Elchalal U, Sharon E, Nokrian M, Ezra Y. External cephalic version for breech presentation with or without spinal analgesia in nulliparous women at term: a randomized controlled trial. Obstet Gynecol. 2007 Dec;110(6):1343-50. doi: 10.1097/01.AOG.0000295605.38175.7b. PMID 18055730

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (6.2) | 28.6 (3.9) | 29.5 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Having Successful Conversion to Cephalic Presentation
Description: Successful conversion of breech fetus to cephalic presentation
Time Frame: Immediately upon completion of the ECV procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
Participants | 3 | 2

2. Secondary Outcome: Cesarean Delivery
Description: Presence of cesarean delivery
Time Frame: Immediately after ECV procedure or during subsequent labor and delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

3. Secondary Outcome: Fetal Presentation at Time of Delivery
Description: Cephalic presentation of the fetus during participant delivery
Time Frame: Labor and Delivery (approximately 12 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
Participants | 3 | 3

4. Secondary Outcome: Cost of ECV Procedure and Hospital Stay (Mother)
Description: Cost of ECV procedure and hospital stay (mother)
Time Frame: ECV procedure and during labor, delivery, and immediate postpartum period (up to 42 days)
Population: Data were not collected for this outcome because of multiple changes to the electronic medical record platforms during the study period and loss of analytics team resources that preclude analysis. There is no possibility of data collection for this secondary outcome.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cost of ECV Procedure and Hospital Stay (Neonate)
Description: Cost of neonate's hospitalization after delivery
Time Frame: Birth to hospital discharge (up to 42 days)
Population: as for outcome 4
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Shoulder Dystocia
Description: Presence of shoulder dystocia during delivery
Time Frame: Labor and Delivery (approximately 12 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

7. Secondary Outcome: Rupture of Membranes
Description: Presence of rupture of membranes after ECV procedure
Time Frame: Within 1 hour of ECV procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

8. Secondary Outcome: Emergency Cesarean Delivery
Description: Need for emergency cesarean delivery during or after ECV procedure
Time Frame: During or within 1 hour of performing ECV procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

9. Secondary Outcome: Pelvic Hematoma
Description: Development of a pelvic hematoma within 1 hour of ECV procedure
Time Frame: During or within 1 hour of performing ECV procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

10. Secondary Outcome: Procedural Pain During Device Insertion
Description: Visual analogue pain score after insertion of balloon device (100mm visual analogue scale where 0 =no pain and 100=extreme pain).
Time Frame: Within 2 minutes after insertion of balloon device.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
units on a scale | 29 [0 to 69] | 59.6 [3 to 85]

11. Secondary Outcome: Number of Attempts
Description: Number of attempted ECV procedures to convert fetus from breech to cephalic presentation
Time Frame: Immediately after ECV procedure
Measure: Mean (Standard Deviation); unit: Number of attempts
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
Number of attempts | 2.3 (1.4) | 2.6 (1.5)

12. Secondary Outcome: Cost of Hospital Stay for ECV Procedure
Description: Total cost of the hospital stay for the ECV procedure
Time Frame: Patient arrival to labor unit for ECV procedure and discharge home (up to 72 hours)
Population: as for outcome 4
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Procedural Pain Prior to Device Insertion.
Description: Baseline visual analogue pain score prior to insertion of balloon device (100mm visual analogue scale where 0 =no pain and 100=extreme pain).
Time Frame: Within 3 minutes prior to insertion of device.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Control: Non-inflation of balloon device
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
units on a scale | 4.8 [0 to 12] | 10.4 [0 to 30]

14. Secondary Outcome: Procedural Pain After Inflation of Device or Sham Inflation.
Description: Visual analogue pain score after inflation or sham inflation of balloon device (100mm visual analogue scale where 0 =no pain and 100=extreme pain).
Time Frame: Within 1 minute after device inflation or sham inflation.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
units on a scale | 22 [0 to 75] | 31 [4 to 60]

15. Secondary Outcome: Pain After External Cephalic Version Attempt.
Description: Visual analogue pain score after ECV procedure (100mm visual analogue scale where 0 =no pain and 100=extreme pain).
Time Frame: Within 2 minutes of ECV procedure completion.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 6 | 5
units on a scale | 38.7 [10 to 60] | 29.2 [0 to 58]

ADVERSE EVENTS:
Time Frame: 1 hour after completion of ECV procedure until discharge after delivery (average of 3.5 weeks)
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT04538261/Prot_SAP_001.pdf